CLINICAL TRIAL: NCT04657133
Title: The Safety and Efficacy of Remote Ischemic Conditioning for the Treatment of Intracerebral Hemorrhage: A Multicenter, Randomized, Controlled Study
Brief Title: Remote Ischemic Conditioning for the Treatment of Intracerebral Hemorrhage
Acronym: RICH-2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RICH-2
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Intracerebral Hemorrhage; Acute Stroke
Keywords: Therapy; Neuroprotection
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Subjects in the intervention group will receive remote ischemic conditioning and standard background medical treatment.
  Interventions: Device: Remote ischemic conditioning; Drug: Standard medication therapy
- Sham group (Placebo Comparator): Subjects in the placebo group will receive sham remote ischemic conditioning and standard background medical treatment alone.
  Interventions: Device: Sham remote ischemic conditioning; Drug: Standard medication therapy

INTERVENTIONS:
Device: Remote ischemic conditioning — RIC is a non-invasive therapy that performed by an electric autocontrol device with cuff placed on arm. RIC procedures consist of five cycles of 5-min inflation (200 mmHg) and 5-min deflation of cuff on one arm. The procedure will be performed once daily for consecutive 7 days after enrollment.
  Other Names: RIC
  Arms: Intervention group
Device: Sham remote ischemic conditioning — Sham RIC will be performed by the same electric autocontrol device with cuff placed on arm. Sham RIC procedures consist of five cycles of 5-min inflation (30 mmHg) and 5-min deflation of cuff on one arm. The procedure will be performed once daily for consecutive 7 days after enrollment.
  Other Names: Sham RIC
  Arms: Sham group
Drug: Standard medication therapy — Standard medication therapy will be performed according to the national and international guidelines.

SUMMARY:
Intracerebral hemorrhage (ICH) results from the rupture of small vessels damaged by chronic hypertension, amyloid angiopathy or other disease. Currently, ICH has been a devastating type of stroke that lacking effective therapy. Remote ischemic conditioning (RIC), a systematically protective strategy, has been found to have neuroprotective effects by in patients with ischemic stroke. In addition, animal studies show that RIC is safe in ICH model and it could accelerate the absorption of hematoma. In a previous clinical study (RICH-1), RIC have been found to be safe and well-tolerated in patients with ICH. Therefore, the investigators plan to undertake this study to further evaluate the safety and efficacy of RIC in patients with ICH.

The investigators hypothesize that treatment with RIC will accelerate the absorption of hematoma and improve patients' functional outcomes. Results of this study can potentially bring into account new means to improve the outcomes of ICH patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 80 years
2. The diagnosis of supratentorial ICH is confirmed by brain CT scan
3. Hematoma volume of 10 to 30 ml and Glasgow Coma Score (GCS)>8 at randomization.
4. National Institutes of Health Stroke Scale (NIHSS)≥6 and ≤20 points at randomization.
5. Randomization and starting treatment between 24 and 48 hours of symptom ictus.
6. Signed and dated informed consent is obtained.

Exclusion Criteria:

1. Planned surgical evacuation of ICH prior to administration of investigational intervention
2. ICH concomitant with subarachnoid hemorrhage or intraventricular hemorrhage
3. Suspected secondary ICH related to tumor, ruptured aneurysm or arteriovenous malformation, hemorrhagic transformation of an ischemic infarct, or venous sinus thrombosis
4. Patients with a pre-existing neurological deficit (mRS>1) or psychiatric disease that would confound the neurological or functional evaluations.
5. Coagulopathy - defined as elevated aPTT or INR >1.3 upon presentation; concurrent use of direct thrombin inhibitors (such as dabigatran), direct factor Xa inhibitors (such as rivaroxaban or apixaban), or low-molecular-weight heparin
6. Severe renal disease (i.e., renal disorder requiring dialysis ) or eGFR <30ml/min/1.73m2
7. Severe liver disorder, or ALT >3 times or bilirubin >2 times upper limit of normal
8. Known severe hearing loss or cognitive impairment
9. Known pregnancy, or positive pregnancy test, or breastfeeding
10. Patients known or suspected of not being able to comply with the study protocol due to alcoholism, noncompliance or any other cause
11. Life expectancy of less than 90 days due to co-morbid conditions
12. Concurrent participation in another research protocol for investigation of another experimental therapy
13. Severe, sustained hypertension (Systolic blood pressure> 180 mmHg or diastolic blood pressure> 110 mmHg).
14. Contraindication for remote ischemic conditioning: severe soft tissue injury, fracture, or peripheral vascular disease in the upper limbs.
15. Any condition which, in the judgement of the investigator, might increase the risk to the patient.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients With Modified Rankin Scale (mRS) Score 0-2 at 90 Days | 0-90 days.
  The mRS ranges from 0 to 6, with higher scores indicating worse outcome. The primary outcome measure is the mRS score, dichotomized to define favorable functional outcome as mRS 0-2 at 90 days.

SECONDARY OUTCOMES:
Proportion of Patients With mRS Score 0-3 at 90 Days | 90 days
  The mRS ranges from 0 to 6, with higher scores indicating worse outcome. Another measure of efficacy is the mRS score, dichotomized to define good functional outcome as mRS 0-3 at 90 days.
Proportion of Patients With mRS Score 0-2 at 180 Days | 180 days
  The mRS ranges from 0 to 6, with higher scores indicating worse outcome. Another measure of efficacy is the mRS score, dichotomized to define good functional outcome as mRS 0-2 at 180 days.
Proportion of Patients With mRS Score 0-3 at 180 Days | 180 days
  The mRS ranges from 0 to 6, with higher scores indicating worse outcome. Another measure of efficacy is the mRS score, dichotomized to define good functional outcome as mRS 0-3 at 180 days.
Number of Subjects Experiencing Serious Adverse Events | 90 days
  Number of subjects experiencing Serious adverse events at any time from randomization through day 90
Number of Subjects With Serious Adverse Events Within 7 Days | 7 days
  Number of Subjects Experiencing Serious Adverse Events within 7 days of randomization

OTHER OUTCOMES:
Changes of intracerebral hematoma volume | 0-7 days after enrollment.
  Intracerebral hematoma volume (ml) is assessed by CT brain scan
Changes of perihematomal edema volume | 0-7 days after enrollment.
  Perihematomal edema volume (ml) is assessed by CT brain scan
Ordinal Distribution of Scores on mRS at Day 90 | 90 days
  The overall ordinal distribution of scores on mRS at 90 days in all subjects of two groups will be determined.
Ordinal Distribution of Scores on mRS at Day 180 | 180 days
  The overall ordinal distribution of scores on mRS at 180 days in all subjects of two groups will be determined.

CONTACTS AND LOCATIONS:
Locations (13):
- China (13):
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Red Cross Emergency Rescue Center, Beijing, Beijing Municipality
  - Beijing Renhe Hospital, Beijing, Beijng
  - Chengde Central Hospital, Chengde, Hebei
  - The Six People's Hospital of Hengshui, Hengshui, Hebei
  - Nanshi Hospital of Nanyang, Nanyang, Henan
  - Tongliao Municipal Hosptial, Tongliao, Inner Mongolia
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality
  - Jiaxing Second Hospital, Jiaxing, Zhejiang
  - Shaoxing People's Hospital, Shaoxing, Zhejiang
  - Zhuji People's Hospital of Zhejaing Province, Zhuji, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shoamanesh A, Patrice Lindsay M, Castellucci LA, Cayley A, Crowther M, de Wit K, English SW, Hoosein S, Huynh T, Kelly M, O'Kelly CJ, Teitelbaum J, Yip S, Dowlatshahi D, Smith EE, Foley N, Pikula A, Mountain A, Gubitz G, Gioia LC. Canadian stroke best practice recommendations: Management of Spontaneous Intracerebral Hemorrhage, 7th Edition Update 2020. Int J Stroke. 2021 Apr;16(3):321-341. doi: 10.1177/1747493020968424. Epub 2020 Nov 11. PMID 33174815
- [Background] Hemphill JC 3rd, Greenberg SM, Anderson CS, Becker K, Bendok BR, Cushman M, Fung GL, Goldstein JN, Macdonald RL, Mitchell PH, Scott PA, Selim MH, Woo D; American Heart Association Stroke Council; Council on Cardiovascular and Stroke Nursing; Council on Clinical Cardiology. Guidelines for the Management of Spontaneous Intracerebral Hemorrhage: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2015 Jul;46(7):2032-60. doi: 10.1161/STR.0000000000000069. Epub 2015 May 28. PMID 26022637
- [Background] Zhao W, Jiang F, Li S, Liu G, Wu C, Wang Y, Ren C, Zhang J, Gu F, Zhang Q, Gao X, Gao Z, Song H, Ma Q, Ding Y, Ji X; RICH-1 Investigators. Safety and efficacy of remote ischemic conditioning for the treatment of intracerebral hemorrhage: A proof-of-concept randomized controlled trial. Int J Stroke. 2022 Apr;17(4):425-433. doi: 10.1177/17474930211006580. Epub 2021 Apr 7. PMID 33739197